CLINICAL TRIAL: NCT03295344
Title: Study of Diaphragm Mobility on Tissue Doppler (Thoracotomy vs Sternotomy in Diaphragm Dysfunction Following Heart Surgery)
Brief Title: Study of Diaphragm Mobility on Tissue Doppler
Acronym: DD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BOUARD ELLOUZE 2016
Record Dates: First submitted 2017-09-25; First posted 2017-09-27 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Heart Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: Diaphragm ultrasonography
- Healthy volunteers
  Interventions: Other: Tissue Doppler

INTERVENTIONS:
Other: Diaphragm ultrasonography — Spontaneously breathing patients in the ½ seated position Heart transducer at the medio axillary position, parallel to the axis of the body, last intervertebral spaces
  US mode:
  2D = Evaluation of the pulmonary parenchyma Time-Movement (TM) = Evaluation of diaphragm muscle shortening in the apposition zone + Evaluation of diaphragm mobility in the posterior 1/3 of the diaphragm dome Tissue Doppler Imaging (TDI) = Evaluation of diaphragm mobility in the diaphragm dome Collection of different daily clinical data
  Groups: Patients
Other: Tissue Doppler — Determine the threshold value for diaphragm mobility
  Groups: Healthy volunteers

SUMMARY:
Diaphragm dysfunction is found in 10 to 90% of patients following heart surgery.

In current practice diaphragm dysfunction is evaluated by 2D ultrasonography. Tissue Doppler is a validated technique to study heart contractility. Its use in the analysis of diaphragm function must be evaluated to determine its interest as a diagnostic tool.

Better understanding of diaphragm dysfunction following heart surgery will lead to earlier management of post-operative respiratory complications and the implementation of preventive pre-operative measures.

We intend to look for correlations between the TM (Time-Movement) mode and tissue Doppler in the assessment of diaphragm mobility.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative period following heart surgery

Exclusion Criteria:

* Patients younger than 18 years old
* Existence of a neuro-muscular disease
* Widened surgical approach
* Refusal of the patient
* Impossibility to see diaphragm movement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the post-operative period following heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Measure diaphragm movement in TM (Time-Movement), in tissue Doppler | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France